CLINICAL TRIAL: NCT04940832
Title: A Single Blinded Randomized Controlled Clinical Trial Comparing Outcome Measures of Pulsed Radiofrequency of the Genicular Nerves When Performed With and Without Concomitant Local Corticosteroid Administration
Brief Title: Outcome Measures of Pulsed Radiofrequency of the Genicular Nerves When Performed With and Without Concomitant Local Corticosteroid Administration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Itay GoorAryeh, Doctor Head of Pain Clinics, Sheba Medical Center, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Knee_pain_radiofrequency
Record Dates: First submitted 2021-06-09; First posted 2021-06-28 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Knee Pain Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- radiofrequency with corticosteroids (Active Comparator): corticosteroids- 80mg depo-medrol Pulsed radiofrequency to 42 derees celsius for 6 minutes
  Interventions: Device: pulsed radiofrequency modulation
- radiofrequency without corticosteroids (Active Comparator): Pulsed radiofrequency to 42 derees celsius for 6 minutes
  Interventions: Device: pulsed radiofrequency modulation

INTERVENTIONS:
Device: pulsed radiofrequency modulation — a percutaneous needle electrode to apply pulsed RF signals that modulate the activity of sensory nerves. The pulsing of the RF signal permits a maximum temperature to be achieved - usually 42 Celsius. This helps prevent collateral damage from occurring during the procedure and should help reduce procedural complications.

SUMMARY:
A single blinded randomized controlled trial to compare outcomes of patients with chronic knee pain receiving radiofrequency with or without corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with pain secondary to osteoarthritis of the knee
* Age of 18 years and up
* Fits criteria for procedure of genicular nerve block and pulsed radiofrequency neuromodulation

Exclusion Criteria:

* Patients who are incapable of judgment and/or to give informed consent
* Patients who are pregnant
* Patients who are under 18 years old
* Patients who have allergies to local anesthetic
* Patients with platelet dysfunction or bleeding disorders
* Patients who are currently mentally unstable
* Patients who have a diagnosis of fibromyalgia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in chronic knee pain | 2nd and 6th week
  Measured by the Knee injury and Osteoarthritis Outcome Score; higher scores indicating that the patients experiences more impairment (All items are scored 0-4; for each subscale the scores are transformed to a 0-100 scale; 0 representing extreme knee problems and 100 representing no knee problems).

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No